CLINICAL TRIAL: NCT04536077
Title: Testing the Immunologic Effects of CDX-301 and CDX-1140 in Resectable Pancreatic Cancer Patients
Brief Title: Immunologic Effects of CDX-301 and CDX-1140 in Resectable Pancreatic Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Celldex decision
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celldex Therapeutics (Industry); The Foundation for Barnes-Jewish Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202011125; 1R01CA262506 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer; Cancer of the Pancreas; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CDX-1140 Monotherapy (Experimental): Patients randomized to the CDX-1140 monotherapy arm will receive a single IV infusion at a dose of 1.5 mg/kg, with surgery to follow 7-12 days after administration of CDX-1140.
  Interventions: Drug: CDX-1140; Procedure: Research blood draw
- CDX-1140 + CDX-301 (Experimental): Patients randomized to the CDX-301 + CDX-1140 arm will receive CDX-301 at 75 mcg/kg/day as a subcutaneous injection every day for 5 days (Days 1-5) with CDX-1140 IV at 1.5 mg/kg on Day 8 +/-1 day. Surgery will be 7-12 days after administration of CDX-1140.
  Interventions: Drug: CDX-301; Drug: CDX-1140; Procedure: Research blood draw

INTERVENTIONS:
Drug: CDX-301 — The drug will be supplied free of charge by Celldex
  Arms: CDX-1140 + CDX-301
Drug: CDX-1140 — The drug will be supplied free of charge by Celldex
Procedure: Research blood draw — At screening; prior to first therapeutic dose of CDX-1140, on the day of the infusion; and at the time of surgery

SUMMARY:
The central hypothesis is that the addition of CDX-301 to CDX-1140 radically improves anti-tumor immunity in patients with pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed surgically resectable pancreatic ductal adenocarcinoma, but not adenosquamous/squamous pancreas cancers (as determined by operating surgeon or tumor board). Patients who have previously received chemotherapy for his/her pancreas cancer within the past 6 months and who are now deemed resectable are also eligible for this trial.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500 /cumm
  * Platelets ≥ 100,000 /cumm
  * Hemoglobin ≥ 9.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance ≤ 1.5 x IULN or glomerular filtration rate of ≥ 60 mL/min
  * INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * Albumin ≥ 3.0mg/dL
* The effects of CDX-301 and CDX-1140 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after the last dose of either study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study or for 3 months after the last dose of either study drug, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Immune deficiencies such as HIV.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Currently receiving any other investigational agents or has received any other investigational agents within 4 weeks or 5 half-lives of the planned first dose of study treatment.
* Receipt of chemotherapy within 2 weeks of planned first dose of study treatment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to CDX-301 or CDX-1140 or other agents used in the study.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (for > 1 month of 10 mg prednisone daily, or equivalent) or any other form of immunosuppressive therapy not routinely associated with chemotherapeutic regimen.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, immunosuppression, autoimmune conditions, or underlying pulmonary disease.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, immunosuppression, autoimmune conditions, or underlying pulmonary disease.
* Has an autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected).
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a known history of active TB (bacillus tuberculosis).
* Major surgery within 28 days prior to the first study treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* History of bone marrow or solid organ transplant.
* Patients with a history of myocardial infarction, cerebral vascular accident, thrombosis or pulmonary embolus within 12 months prior to the first dose of study treatment are excluded from this study.
* Patients with known mutations/amplifications in Flt3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roheena Z Panni, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CDX-1140 Monotherapy | CDX-1140 + CDX-301
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Did not start treatment due to surgery needing to occur urgently | 1 | 0
Not completed — Did not start treatment due to disease progression and no longer having resectable disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDX-1140 Monotherapy | CDX-1140 + CDX-301 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Median (Full Range); unit: years] | 69 [53 to 77] | 64 [51 to 74] | 65 [51 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 6 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Amount of Intratumoral Conventional Dendritic Cells (cDCs)
Time Frame: At time of surgery (estimated to be between day 8 and day 20)
Population: Participants were not included in the overall number of participants analyzed if there was insufficient tumor for additional analysis or small tumor size.
Measure: Mean (Standard Deviation); unit: percentage of total cells
Arm/Group | CDX-1140 Monotherapy | CDX-1140 + CDX-301
Number analyzed (Participants) | 4 | 4
percentage of total cells | 0.9615 (0.3699) | 2.631 (0.8024)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through time of surgery (or 60 days after end of treatment if surgery doesn't take place).
Description: If patients did not start treatment with CDX-1140 monotherapy or CDX-1140 + CDX-301 treatment then adverse events were not collected. There was one participant in each arm who did not start treatment, therefore, adverse events were not collected on those two patients.
Arm/Group | CDX-1140 Monotherapy | CDX-1140 + CDX-301
All-Cause Mortality (participants affected / at risk) | 2/8 | 3/8
Serious Adverse Events (participants affected / at risk) | 1/7 | 3/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDX-1140 Monotherapy (N=7) | CDX-1140 + CDX-301 (N=7)
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Flu like symptoms (General disorders) | 1 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDX-1140 Monotherapy (N=7) | CDX-1140 + CDX-301 (N=7)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1
Mouth sores - lower lip (General disorders) | 1 | 0
Chills (General disorders) | 2 | 3
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 3
Fever (General disorders) | 2 | 3
Malaise (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3
Lymphocyte count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Joint inflammation ankles (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint inflammation bilateral hands (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Red rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Flu like symptoms (General disorders) | 0 | 1
Thrush (Infections and infestations) | 0 | 1
Immature granulocyte increased (Investigations) | 0 | 1
Monocyte increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04536077/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT04536077/ICF_001.pdf